CLINICAL TRIAL: NCT01471847
Title: A Phase Ib/Randomized Phase II Study of BEZ235 and Trastuzumab Versus Lapatinib and Capecitabine in Patients With HER2-positive Locally Advanced or Metastatic Breast Cancer Who Failed Prior to Trastuzumab
Brief Title: A Phase Ib/II Study of BEZ235 and Trastuzumab in Patients With HER2-positive Breast Cancer Who Failed Prior to Trastuzumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235B2203
Record Dates: First submitted 2011-10-10; First posted 2011-11-16 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2018-02

CONDITIONS: Locally Advance Breast Cancer (LABC); Metastatic Breast Cancer (MBC)
Keywords: Locally advanced; metastatic; breast cancer; HER2 positive; PI3K; mTOR; trastuzumab; targeted therapy; LABC; MBC
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — dactolisib; Lapatinib; Capecitabine; Clinical Trials, Phase II as Topic

ARMS (2):
- BEZ235 + Trastuzumab (Phase l /Phase ll) (Experimental): Phase l: Eligible patients will receive increasing doses of oral BEZ235 administered on a continuous twice daily (BID) schedule + weekly trastuzumab at a fixed dose of 2 mg/kg. Treatment will be organized into cycles of 28 days.
  Phase ll: Eligible patients will receive weekly trastuzumab (2 mg/kg) + oral BEZ235 on a continuous twice daily (BID schedule) at the MTD or RP2D.
  Treatment will be organized into cycles of 21 days.
  Interventions: Drug: BEZ235 + Trastuzumab Phase l/Phase ll)
- Lapatinib + Capecitabine (Phase II) (Active Comparator): Eligible patients will receive lapatinib (1250 mg given orally once daily on days 1 through 21) in combination with capecitabine (2000 mg/m2/day administered orally in 2 doses approximately 12 hours apart on days 1 through 14). Treatment will be organized into cycles of 21 days .
  Interventions: Drug: Lapatinib + Capecitabine (Phase II)

INTERVENTIONS:
Drug: BEZ235 + Trastuzumab Phase l/Phase ll) — Phase l: Patients will receive increasing doses of oral BEZ235 (BID) together with standard weekly trastuzumab at a fixed dose. BEZ235 doses will be escalated in cohorts of 3 to 6 patients guided by an adaptive Bayesian logistic regression model with overdose control until MTD/RP2D has been established.
  Phase ll: If randomized to the trastuzumab + BEZ235 arm, patients will receive standard weekly trastuzumab in combination with oral BEZ235 (BID) at the MTD or RP2D and will continue on study treatment until PD, unacceptable toxicity or until other pre-defined discontinuation criteria are met. They will have regular safety assessments and will be evaluated for response to treatment according to RECIST every 2 cycles for the first 36 weeks then every 12 weeks until disease progression (or start of new anti-neoplastic therapy).
  Arms: BEZ235 + Trastuzumab (Phase l /Phase ll)
Drug: Lapatinib + Capecitabine (Phase II) — If randomized to the lapatinib + capecitabine treatment arm, patients will receive standard lapatinib plus capecitabine until PD, unacceptable toxicity or until other pre-defined discontinuation criteria are met.
  Patients will have regular safety assessments and will be evaluated for response to treatment according to RECIST every 2 cycles for the first 36 weeks then every 12 weeks until disease progression (or start of new anti-neoplastic therapy). After progression, survival f-up will continue.
  All patients participating in the Phase II part of the study will be required to have available archival or fresh tumor tissue for biomarker analysis prior to treatment start
  Arms: Lapatinib + Capecitabine (Phase II)

SUMMARY:
This is a prospective, multi-center, open-label, phase Ib/ II study (two parts) with patients that have locally advanced or metastatic HER2+ breast cancer. The first part (phase Ib) will investigate the MTD/ RP2D of the combination therapy of BEZ235 BID and weekly trastuzumab using a Bayesian model. Once MTD/ RP2D is established the second part (phase II) will start. Phase II will evaluate the efficacy and the safety of weekly trastuzumab plus BEZ235 BID compared to capecitabine and lapatinib.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a female ≥ 18 years of age
* Patient has a histologically and/or cytologically confirmed diagnosis of HER2-positive invasive breast cancer with inoperable locally advanced or metastatic disease
* Patients with controlled or asymptomatic CNS metastases are eligible
* Patient has adequate bone marrow and organ functions, and has recovery from all clinically significant toxicities related to prior anti-neoplastic therapies
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelets ≥ 100 x 109/L
* Hemoglobin (Hgb) ≥ 9.0 g/dL
* INR ≤ 2
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN (or ≤ 5.0 x ULN if liver metastases are present)
* Total serum bilirubin ≤ 1.5 x ULN (in patients with known Gilbert Syndrome, a total bilirubin ≤ 3.0 x ULN, with direct bilirubin ≤ 1.5 x ULN)
* Serum creatinine ≤ 1.5 x ULN
* Fasting plasma glucose (FPG) ≤ 140mg/dL [7.8 mmol/L]
* HbA1c ≤ 8%
* Patient has received prior trastuzumab (alone or in combination) but NO more than 3 prior cytotoxic chemotherapy lines
* Prior endocrine and radiotherapy allowed
* Patient has ECOG performance status of 0-2 (Phase Ib) or 0-1 (Phase II)

Additional inclusion criteria for phase II:

* Available tumor tissue (archival or fresh) for biomarker analysis; known PI3K activation status
* At least one measurable lesion as per RECIST 1.1
* Patient has received prior treatment with a taxane
* Patient has "trastuzumab-resistance disease" defined as:
* Recurrence while on trastuzumab (or T-DM1) or within 12 months since the last infusion in the adjuvant setting
* Progression while on or within 4 weeks since the last infusion of trastuzumab (or T-DM1) in the locally advanced or metastatic setting

Exclusion Criteria:

* Previous treatment with PI3K and/or mTOR inhibitors
* Symptomatic/uncontrolled Central Nervous System (CNS) metastases
* Concurrent malignancy or malignancy in the last 3 years prior to enrollment
* Wide field radiotherapy ≤ 28 days or limited field radiation for palliation ≤ 14 days prior to starting study drug
* Active cardiac disease (e.g. LVEF less than institutional lower limit of normal, QTcF > 480 msec, unstable angina pectoris, ventricular, supraventricular or nodal arrhythmias)
* Inadequately controlled hypertension
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BEZ235
* Treatment at start of study treatment with drugs with a known risk to induce Torsades de Pointes, moderate and strong inhibitors or inducers of isoenzyme CYP3A4, warfarin and coumadin analogues, LHRH agonists
* Intolerance or contraindications to trastuzumab treatment
* Pregnant or nursing (lactating) woman

Additional exclusion criteria for phase II:

* Prior treatment with capecitabine and lapatinib
* Intolerance or contraindications to capecitabine and lapatinib
* Previous treatment with HER-2 targeted agents other than trastuzumab or T-DM1
* Peripheral neuropathy ≥ Grade 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) in the first cycle - phase lb | First treatment cycle (28 days)
  DLT is defined as treatment-related toxicity (classified according Common Toxicity Criteria for Adverse Events (CTCAE) Version 4) occurring during the first 28 treatment days and meeting specific protocol-predefined criteria.
  The information will be integrated in a Bayesian logistic regression model with overdose control to estimate the maximum tolerated dose (MTD)
Progression Free Survival (PFS) based on local radiological assessment - phase ll | Randomization, disease progression or start of of new anti-neoplastic therapy (expected average: 12 months)
  PFS is defined as the time from randomization until objective tumor progression or death from any cause. Radiological assessments will be performed every 6 weeks for the first 36 weeks after treatment start, then every 12 weeks.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) - Phase lb | Randomization, Randomization, disease progression or start of of new anti-neoplastic therapy (expected average: 12 months)
  Time from treatment start until objective tumor progression or death from any cause. Radiological assessments will be performed every 8 weeks for the first 32 weeks after treatment start, then every 12 weeks.
Overall Response Rate (ORR)- Phase lb | 12 months
  Proportion of patients with a best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1
Clinical Benefit Rate (CBR) (Phase lb) | 12 months
  Proportion of patients with a best overall response of CR, PR or stable disease (SD) with a duration of 24 weeks or longer according to RECIST 1.1
Frequency and severity of Adverse Events - Phase lb | until 30 days after treatment discontinuation
  Incidence of adverse events (based on common terminology criteria for adverse events (CTCAE) Version 4) summarized by system organ class and/or preferred term, severity and relation to study treatment.
BEZ235 plasma and trastuzumab serum concentrations - phase lb | Pre-dose (cycle 1 through 9) and 4-6 hours post-dose (cycle 1 and 2)
  BEZ235 plasma and trastuzumab serum concentrations obtained during the two sampling windows (pre-dose and post-dose). No pharmacokinetic parameters will be calculated and no formal statistical analysis will be performed.
Overall Response Rate (ORR) - phase ll | 12 months
  Proportion of patients with a best overall response of CR or PR according to RECIST 1.1
Clinical Benefit Rate (CBR) - phase ll | 12 months
  Proportion of patients with a best overall response of CR, PR or SD with a duration of 24 weeks or longer according to RECIST 1.1
Time to overall response (TTR) - phase ll | 12 months
  Time from randomization until first documented response.
Duration of overall response (DR) - phase ll | 12 months
  Time between the first documented response and first documented progression or death due to underlying cancer.
Median overall survival (OS) (phase ll) | Randomization, death (expected average:24 months)
  Time from randomization to the date of death due to any cause.
PFS based on central radiological assessment (phase ll) | Randomization, disease progression or start of of new anti-neoplastic therapy (expected average: 12 months)
  Time from randomization until objective tumor progression or death from any cause. Radiological assessments will be performed every 6 weeks for the first 36 weeks after treatment start, then every 12 weeks, centrally collected and read.
Frequency and severity of adverse events (phase ll) | Until 30 days after treatment discontinuation
  Incidence of adverse events (based on CTCAE Version 4) summarized by system organ class and/or preferred term, severity and relation to study treatment.
Efficacy in subgroups of patients with activated/non-activated PI3K pathway (phase ll) | 12 months
  Efficacy (e.g. PFS, ORR, CBR) according to PI3K activation and treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Madrid, Spain
- United Kingdom (2):
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Manchester

REFERENCES:
- See also: Results for CBEZ235B2203 can be found on the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8603